CLINICAL TRIAL: NCT06180044
Title: Quantification of Physiologic Burden to the Surgeon During Orthopaedic Surgery
Brief Title: Physiologic Burden to the Surgeon During Orthopaedic Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Pelt, Principle Investigator, University of Utah
Other Study IDs: 170873
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Physiological Stress
Keywords: Surgeon; Orthopaedic surgery; Hexoskin Smart Vest; Physiologic data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator's plan to quantify the physiologic impact of orthopaedic surgery on the surgeon and operating team.

DETAILED DESCRIPTION:
The prevalence of musculoskeletal pain among orthopaedic surgeons is inordinately high. Poor surgical ergonomics and physiological stress have been shown to impair surgical performance and cause injuries. Various approaches, techniques and instruments have been designed to improve surgical outcomes for patients. There has been nominal research in the area of occupational hazards such surgeries impose upon the surgeon. Several studies have demonstrated a higher risk of cervical spondylosis and rotator cuff tears amongst surgeons. However, little has been studied on the impacts of some of these approaches, techniques, and instruments on surgeons' physiologic measures.

The investigator's will use The Hexoskin Smart Vest to capture physiological data from surgeons during the study.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic surgeons, orthaopedic fellows, and orthopaedic residents.
* Up to 750 surgical patients of the participating surgeons will be included for demographic chart review.

Exclusion Criteria:

* Non-surgeons, fellows, or residents.
* Female participants that are or become pregnant.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Orthopaedic surgeons, orthopaedic fellows, and orthopaedic residents performing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Average Heart Rate (beats per minute, bpm) | 30 minutes before surgery
  Average surgeon heart rate prior to surgery.
Average Heart Rate (beats per minute, bpm) | During entire surgical procedure
  Average surgeon heart rate during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pelt, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States